CLINICAL TRIAL: NCT04106843
Title: A Phase II Study to Evaluate the Effects of 177Lu-DOTATATE in Patients With Unresectable and Progressive Rare Metastatic Endocrine Carcinomas: Medullary Thyroid Cancer, Parathyroid Carcinoma, Pituitary Carcinoma, and Malignant Pheochromocytoma/Paraganglioma
Brief Title: Radioactive Drug (177Lu-DOTATATE) for the Treatment of Locally Advanced, Metastatic, or Unresectable Rare Endocrine Cancers
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No Participants Registered
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-0947; NCI-2019-05859 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0947 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-09-25; First posted 2019-09-27 (Actual); Last update posted 2020-09-07 (Actual); Status verified 2020-09

CONDITIONS: Locally Advanced Adrenal Gland Pheochromocytoma; Locally Advanced Paraganglioma; Metastatic Adrenal Gland Pheochromocytoma; Metastatic Paraganglioma; Metastatic Parathyroid Gland Carcinoma; Pituitary Gland Carcinoma; Somatostatin Receptor Positive; Stage III Thyroid Gland Medullary Carcinoma AJCC v8; Stage IV Thyroid Gland Medullary Carcinoma AJCC v8; Stage IVA Thyroid Gland Medullary Carcinoma AJCC v8; Stage IVB Thyroid Gland Medullary Carcinoma AJCC v8; Stage IVC Thyroid Gland Medullary Carcinoma AJCC v8; Unresectable Adrenal Gland Pheochromocytoma; Unresectable Paraganglioma
MeSH Terms: conditions — Pheochromocytoma; Paraganglioma; Parathyroid Neoplasms; Pituitary Neoplasms; Carcinoma, Medullary | interventions — lutetium Lu 177 dotatate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (177Lu-DOTATATE) (Experimental): Patients receive 177Lu-DOTATATE IV over 30 minutes every 8-16 weeks. Treatment continues for up to 52 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Lutetium Lu 177 Dotatate

INTERVENTIONS:
Drug: Lutetium Lu 177 Dotatate — Given IV
  Other Names: 177 Lu-DOTA-TATE; 177 Lu-DOTA-Tyr3-Octreotate; 177Lu-DOTA0-Tyr3-Octreotate; Lutathera; Lutetium Lu 177 DOTA(0)-Tyr(3)-Octreotate; Lutetium Lu 177-DOTA-Tyr3-Octreotate; lutetium Lu 177-DOTATATE; Lutetium Oxodotreotide Lu-177

SUMMARY:
This phase II trial studies how well 177Lu-DOTATATE works in treating patients with rare endocrine cancers that have spread from where they started to nearby tissue or lymph nodes (locally advanced), spread to other places in the body (metastatic), or cannot be removed by surgery (unresectable). Radioactive drugs, such as 177Lu-DOTATATE, may carry radiation directly to cancer cells and not harm normal cells. 177Lu-DOTATATE may help to control endocrine cancers compared to standard treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Objective response rate (ORR) by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 determined by Ia. Computed tomography (CT) or Ib. Magnetic resonance imaging (MRI).

SECONDARY OBJECTIVES:

I. To estimate progression-free survival at 1-year. II. To correlate blood pressure control and change/discontinuation of antihypertensive medications with tumor responses in patients with pheochromocytomas and paragangliomas (PHPGs).

III. To correlate plasma metanephrines and chromogranin A with tumor responses in patients with PHPGs.

IV. To correlate calcitonin, carcinoembryonic antigen, and chromogranin A with tumor responses in patients with medullary thyroid carcinoma (MTCs).

V. To correlate pituitary hormones (depending on particular tumor, e.g. prolactin for prolactinomas, insulin-like growth factor (IGF-1) for acromegaly, adrenocorticotropic hormone (ACTH) and 24-hour urine free cortisol for Cushing disease, and chromogranin A with tumor responses in patients with functional pituitary carcinomas).

VI. To correlate calcium, intact parathyroid hormone (iPTH), and chromogranin A with tumor responses in patients with parathyroid carcinoma.

VII. Toxicity assessment by the Common Terminology Criteria for Adverse Events version 5.0 (CTCAE 5.0).

VIII. To correlate tumor responses with tumor uptake score in somatostatin receptor scintigraphy, overall prognosis and responsiveness to lutetium Lu 177 dotatate (177Lu-DOTATATE).

IX. To determine the percentage of tumors that demonstrate uptake on diagnostic 68Gallium-DOTATATE positron emission tomography (PET)/CT that would make treatment with 177Lu-DOTATATE feasible.

EXPLORATORY OBJECTIVES:

I. To evaluate pituitary function in all patients to look for possible radiation late effects on the pituitary gland.

II. To estimate best biochemical response for specific tumor markers in patients with non-measurable disease.

III. To correlate biochemical response in patients with non-measurable disease with RECIST 1.1 tumor response criteria for patients with non-measurable disease.

OUTLINE:

Patients receive 177Lu-DOTATATE intravenously (IV) over 30 minutes every 8-16 weeks. Treatment continues for up to 52 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at week 72 and then every 24 weeks for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of PHPG, MTC, parathyroid or pituitary tumor
* Locally advanced or distantly metastatic disease not amenable to surgery
* Patients should have somatostatin receptor (SSTR)+ tumor as determined by 68Ga-DOTATATE PET/CT imaging. A measurable SSTR+ tumor is defined as having greater than or equal to 10 mm in diameter with uptake higher than or equal to liver and is qualitatively higher and distinguishable from background activity
* In patients with multiple lesions (more than one) as determined by staging CT or MRI, the number of SSTR+ lesions should be more than or equal to the number of SSTR- lesions
* Patients enrolled in cohorts 1-4 should have measurable disease defined by RECIST 1.1
* Patients enrolled in cohort 5 should have non-measurable disease as defined by RECIST 1.1
* Progressive disease per RECIST 1.1 as determined by the investigator within the 12 months preceding study enrollment
* Radiographic assessment of all known disease sites, e.g., by computerized tomography (CT) scan, magnetic resonance imaging (MRI), bone scan as appropriate within 28 days before the first dose of (177)Lu-DOTATATE
* Disease specific hormonal studies to assess abnormal hormonal secretion within 28 days before the first dose of (177)Lu-DOTATATE. These studies may include the following: plasma metanephrines and catecholamines for PHPG, calcitonin and CEA for MTC, prolactin for malignant prolactinomas, IGF-1 for growth hormone secreting malignant somatotropinomas, ACTH for malignant corticotropinomas, intact parathyroid hormone for parathyroid carcinomas
* Eastern Cooperative Oncology Group (ECOG) performance status of =< 2
* Life expectancy of at least 6 months
* Absolute neutrophil count (ANC) >= 1500/mm^3 without colony stimulating factor support (within 4 days prior to the first dose of [177]Lu-DOTATATE)
* Platelets >= 100,000/mm^3 (within 4 days prior to the first dose of [177]Lu-DOTATATE)
* Hemoglobin >= 9 g/dL (within 4 days prior to the first dose of [177]Lu-DOTATATE)
* Bilirubin =< 1.5 x the upper limit of normal (ULN) (within 4 days prior to the first dose of [177]Lu-DOTATATE). For subjects with known Gilbert's disease, bilirubin =< 3.0 mg/dL
* Serum albumin >= 2.8 g/dl (within 4 days prior to the first dose of [177]Lu-DOTATATE)
* Serum creatinine =< 1.5 x ULN or creatinine clearance (CrCl) >= 50 mL/min (within 4 days prior to the first dose of [177]Lu-DOTATATE). For creatinine clearance estimation, the Cockcroft and Gault equation should be used
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 3.0 x ULN (within 4 days prior to the first dose of [177]Lu-DOTATATE)
* Random urine protein/creatinine ratio (UPCR) =< 1 (within 4 days prior to the first dose of [177]Lu-DOTATATE)
* Serum phosphorus, calcium, magnesium and potassium >= lower limit of normal (LLN) (within 4 days prior to the first dose of [177]Lu-DOTATATE)
* Capable of understanding and complying with the protocol requirements and has signed the informed consent document
* Sexually active patients (men and women) must agree to use medically accepted barrier methods of contraception (e.g., male or female condom) during the course of the study and for 4 months after the last dose of study drug(s), even if oral contraceptives are also used. All subjects of reproductive potential must agree to use both a barrier method and a second method of birth control during the course of the study and for 6 months after the last dose of study drug(s)
* Women of childbearing potential must have a negative pregnancy test at screening. Women of childbearing potential include women who have experienced menarche and who have not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or are not postmenopausal. Postmenopause is defined as amenorrhea >= 12 consecutive months. Note: women who have been amenorrheic for 12 or more months are still considered to be of childbearing potential if the amenorrhea is possibly due to prior chemotherapy, antiestrogens, ovarian suppression or any other reversible reason

Exclusion Criteria:

* Received cytotoxic chemotherapy (including investigational cytotoxic chemotherapy) or biologic agents (e.g., somatostatin analogues, cytokines or antibodies) within 12 weeks, or nitrosoureas/mitomycin C within 6 weeks before the first dose of study treatment. For patients with acromegaly, Cushing disease, and thyroid-stimulating hormone (TSH) secreting pituitary carcinomas treatment with somatostatin analogues is allowed
* Prior treatment with (177)Lu-DOTATATE or other radionuclide agents (e.g. (131)I meta-iodobenzylguanidine, (131)I Ultratrace Iobenguane)
* Radiation therapy for bone metastasis within 2 weeks, any other external radiation therapy within 4 weeks before the first dose of study treatment. Subjects with clinically relevant ongoing complications from prior radiation therapy are not eligible
* Prior treatment of any small molecule kinase inhibitor (including investigational kinase inhibitor) within 14 days before the first dose of study treatment
* Receipt of any other type of investigational agent within 28 days before the first dose of study treatment
* The subject has not recovered to baseline or CTCAE =< grade 1 from toxicity due to all prior therapies except alopecia and other non-clinically significant adverse events (AEs)
* Prothrombin time (PT)/international normalized ratio (INR) or partial thromboplastin time (PTT) test >= 1.3 x the laboratory ULN within 7 days before the first dose of study treatment
* Uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:

  * Cardiovascular disorders including

    * Congestive heart failure (CHF): New York Heart Association (NYHA) class III (moderate) or class IV (severe) at the time of screening
    * Concurrent uncontrolled hypertension defined as sustained blood pressure (BP) > 150 mm Hg systolic, or > 90 mm Hg diastolic despite optimal antihypertensive treatment within 7 days of the first dose of study treatment
  * Any of the following within 6 months before the first dose of study treatment:

    * Unstable angina pectoris
    * Clinically-significant cardiac arrhythmias
    * Stroke (including transient ischemic attack (TIA), or other ischemic event)
    * Myocardial infarction
* Other clinically significant disorders such as:

  * Active infection requiring systemic treatment within 28 days before the first dose of study treatment
  * Serious non-healing wound/ulcer/bone fracture within 28 days before the first dose of study treatment
  * History of organ transplant
  * Concurrent uncompensated hypothyroidism or thyroid dysfunction within 7 days before the first dose of study treatment; in patients with central hypothyroidism due to pituitary cancer FT4 should be within normal limits, TSH is not evaluable for this cohort
  * Major surgery within 12 weeks before the first dose of study treatment. Complete wound healing from major surgery must have occurred 1 month before the first dose of study treatment. Minor surgery within 28 days before the first dose of study treatment with complete wound healing at least 10 days before the first dose of study treatment. Subjects with clinically relevant ongoing complications from prior surgery are not eligible
* Pregnant or breastfeeding
* A previously identified allergy or hypersensitivity to components of the study treatment formulation
* Unable or unwilling to abide by the study protocol or cooperate fully with the investigator or designee
* Evidence within 2 years of the start of study treatment of another malignancy that required systemic treatment except for cured non-melanoma skin cancer, cured in situ cervical carcinoma, or papillary microcarcinoma as long as there is no evidence of disease
* Any other severe acute or chronic medical or psychiatric condition or laboratory abnormality which, in the judgment of the investigator, would have made the patient inappropriate for entry into this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-06-13 (Estimated); Primary Completion 2020-09-03 (Actual); Study Completion 2020-09-03 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to 52 weeks
  Assessed by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 determined by computed tomography (CT) or magnetic resonance imaging (MRI). Will be calculated as the proportion of patients with complete responses (CR), partial responses (PR), or stable disease (SD) at the CT/MRI assessment time point.

CONTACTS AND LOCATIONS:
Overall Officials: Camilo Jimenez, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org